CLINICAL TRIAL: NCT02170805
Title: Bioavailability of BIBR 953 ZW After Single Oral Doses of Two Different 50 mg Capsules of BIBR 1048 MS With and Without Coadministration of Pantoprazole to Healthy Subjects Relative to Solution. Two Groups, 3-way Crossover, Randomised, Open Trial
Brief Title: Bioavailability of BIBR 1048 MS Single Doses With or Without Pantoprazole in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.17
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Solutions; Pantoprazole

ARMS (2):
- Substudy 1 (Experimental): Three treatments of single administrations of BIBR 1048 MS 50 mg with or without pantoprazole; randomised sequence
  1. BIBR 1048 MS capsule formulation A without pantoprazole;
  2. BIBR 1048 MS capsule formulation A with coadministration of 40 mg pantoprazole (bid);
  3. BIBR 1048 MS powder plus solution without pantoprazole
  Interventions: Drug: BIBR 1048 MS capsule formulation A; Drug: BIBR 1048 MS powder plus solution; Drug: Pantoprazole
- Substudy 2 (Experimental): Three treatments of single administrations of BIBR 1048 MS 50 mg with or without pantoprazole; randomised sequence
  1. BIBR 1048 MS capsule formulation B without pantoprazole;
  2. BIBR 1048 MS capsule formulation B with coadministration of 40 mg pantoprazole (bid);
  3. BIBR 1048 MS powder plus solution without pantoprazole
  Interventions: Drug: BIBR 1048 MS capsule formulation B; Drug: BIBR 1048 MS powder plus solution; Drug: Pantoprazole

INTERVENTIONS:
Drug: BIBR 1048 MS capsule formulation A — BIBR 1048 MS, formulation A 50 mg
  Arms: Substudy 1
Drug: BIBR 1048 MS capsule formulation B — BIBR 1048 MS, formulation B 50 mg
  Arms: Substudy 2
Drug: BIBR 1048 MS powder plus solution — BIBR 1048 MS, powder plus solution 50 mg
Drug: Pantoprazole — Pantoprazole 40 mg
  Other Names: Pantozol®

SUMMARY:
The pharmacokinetics of 50 mg BIBR 1048 administered as two newly developed capsule formulation using melt extrusion technology was assessed in two separate, single dose, 3-way crossover, open design, randomised studies. The 3-way crossover treatments included administration of the tartaric acid solution of 50 mg BIBR 1048, the capsule formulation A or B and administration of the capsules with coadministration of pantoprazole.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with GCP and local legislation
* Age ≥ 18 and ≤ 55 years
* Broca ≥ - 20% and ≤ + 20%

Exclusion Criteria:

* Any findings of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* History or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* History of orthostatic hypotension, fainting spells and blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Any bleeding disorder including prolonged or habitual bleeding
* Other hematologic disease
* Cerebral bleeding (e.g. after a car accident)
* Commotio cerebri
* Intake of drugs with a long half-life (>24 hours) within 1 month prior to administration
* Use of any drugs which might influence the results of the trial within 10 days prior to administration or during trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range
* History of any familial bleeding disorder
* Thrombocytes < 150000/µl

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2001-04; Primary Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (Area under the concentration-time curve the time interval from 0 extrapolated to infinity) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration of study drug
AUC0-tf (Area under the concentration-time curve over the time interval from 0 to the time of the last quantifiable concentration) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration of study drug

SECONDARY OUTCOMES:
Cmax (Maximum measured concentration) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration of study drug
tmax (Time from dosing to the maximum concentration) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration of study drug
t1/2 (Terminal half-life) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration of study drug
MRTtot (Total mean residence time) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration of study drug
CLtot/F (Total apparent clearance) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration of study drug
Vz/F (Apparent volume of distribution) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration of study drug
λz (terminal elimination rate constant) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration of study drug
Changes in aPTT (activated partial thromboplastin time) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration of study drug
Changes in PT (prothrombin time) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration of study drug